CLINICAL TRIAL: NCT04379453
Title: Robot Assisted Percutaneous Cardiovascular Intervention as a Strategy to Reduce or Risk of Intra-Procedure Contamination by COVID-19 and Other Respiratory Viruses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4094-20
Record Dates: First submitted 2020-04-27; First posted 2020-05-07 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-04

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Robot Assisted Percutaneous Cardiovascular Intervention; COVID-19
MeSH Terms: conditions — Coronary Artery Disease; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Robot Assisted Percutaneous Cardiovascular Intervention (Experimental): Robot Assisted Percutaneous Cardiovascular Intervention as a Strategy to Reduce or Risk of Intra-Procedure Contamination by COVID-19 and Other Respiratory Viruses
  Interventions: Procedure: Robot Assisted Percutaneous Cardiovascular Intervention

INTERVENTIONS:
Procedure: Robot Assisted Percutaneous Cardiovascular Intervention — Robot Assisted Percutaneous Cardiovascular Intervention

SUMMARY:
Percutaneous cardiovascular intervention procedures (e.g. coronary angioplasty, peripheral artery angioplasty) must be performed in person, requiring the physical presence of one or more medical, nursing and technical professionals. The control of catheters and interventional materials is performed manually, with the operator positioned next to the patient. This context results in potential for reciprocal exposure to exhaled air, both for the professionals involved and for the patient, with an inherent risk of aerial contamination. It is important to note that interventional procedures are often performed on an urgent or emergency basis (e.g. myocardial infarction), without the possibility of postponement or postponement.

The recent robot-assisted cardiovascular intervention makes it possible to modify this scenario by allowing the procedure to be performed effectively and safely in a position far from the patient. In an environment with high potential for contamination, mainly related to the current pandemic caused by the COVID-19 virus, may prove to be a tactic to expand hospital security.

It is in this sense that the present pilot proposal is inserted, which, ultimately, aims to evaluate the potential of robotic intervention as a strategy to reduce exposure to exhaled air of patients and professionals during the intervention procedure.

DETAILED DESCRIPTION:
Percutaneous cardiovascular intervention procedures (e.g. coronary angioplasty, peripheral artery angioplasty) must be performed in person, requiring the physical presence of one or more medical, nursing and technical professionals. The control of catheters and interventional materials is performed manually, with the operator positioned next to the patient. This context results in potential for reciprocal exposure to exhaled air, both for the professionals involved and for the patient, with an inherent risk of aerial contamination. It is important to note that interventional procedures are often performed on an urgent or emergency basis (e.g. myocardial infarction), without the possibility of postponement or postponement.

The recent robot-assisted cardiovascular intervention makes it possible to modify this scenario by allowing the procedure to be performed effectively and safely in a position far from the patient. In an environment with high potential for contamination, mainly related to the current pandemic caused by the COVID-19 virus, may prove to be a tactic to expand hospital security.

It is in this sense that the present pilot proposal is inserted, which, ultimately, aims to evaluate the potential of robotic intervention as a strategy to reduce exposure to exhaled air of patients and professionals during the intervention procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age> = 18 years;
* Cardiovascular disease characterized by:
* Symptomatic ischemic heart disease and / or objective evidence of myocardial ischemia with one or more target lesions OR
* Symptomatic peripheral arterial disease and / or with objective evidence of the need for percutaneous intervention of one or more target lesions;
* The target lesion (s) must be obstructive and / or aneurysmatic (visual analysis);
* Interventionist planning for all target lesions should include robotic manipulation in at least one treatment period, according to the operator's judgment;
* The patient will be informed about the nature of the study, agree with its rules and will provide written informed consent, approved by the local Ethics Committee.

Exclusion Criteria:

* Platelet count <50,000 cells / mm3 or> 700,000 cells / mm3;
* Total leukometry <3,000 cells / mm3;
* Suspected or documented active liver disease, with blood dyscrasia with INR <1.5;
* Heart transplant recipient;
* Allergies known to aspirin, clopidogrel, ticlopidine, ticagrelor, prasugrel, heparin, antiproliferative agents of the limus family, or stainless steel;
* Patient with a life expectancy of less than 1 month;
* Any significant medical condition that in the investigator's opinion may interfere with the patient's ideal participation in this study;
* Participation in another research in the last 12 months, unless there can be direct benefit to the research subject;
* Any invasive cardiac or non-cardiac treatment scheduled in the first month after the index procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-04-27 (Estimated); Primary Completion 2020-04-27 (Estimated); Study Completion 2020-04-27 (Estimated)

PRIMARY OUTCOMES:
Successful cardiovascular intervention | Until the end of the procedure
  (arterial dilation with residual lesion <50% at angiography and normal anterograde flow)
Performed with the professional team positioned at> 2 meters from the patient for at least 50% of the duration of the intervention | Until the end of the procedure
absence of fatal complications caused by the procedure or acute non-fatal vessel occlusion during index admission | Until the end of the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Lemos, MD, Principal Investigator — Hospital Israelita Albert Einstein
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lemos PA, Franken M, Mariani J Jr, Pitta FG, Oliveira FA, Cunha-Lima G, Caixeta AM, Almeida BO, Garcia RG. Use of robotic assistance to reduce proximity and air-sharing during percutaneous cardiovascular intervention. Future Cardiol. 2021 Aug;17(5):865-873. doi: 10.2217/fca-2021-0024. Epub 2021 Apr 9. PMID 33834847